CLINICAL TRIAL: NCT02027779
Title: An Open Label Safety and Efficacy Extension Study of GreenGene™ F in Previously Treated Patients Diagnosed With Severe Hemophilia A
Brief Title: Safety and Efficacy Extension Study of GreenGene™ F in Previously Treated Patients Diagnosed With Severe Hemophilia A
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Green Cross Corporation (Industry)
Collaborators: Atlantic Research Group (Other)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GreenGene™ F_E_P3
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Hemophilia A
Keywords: GreenGene™ F, Previously Treated Patients
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prophylaxis safety and efficacy substudy (Experimental): Hemostatic efficacy of GreenGene™ F will be assessed by its effectiveness in controlling spontaneous or traumatic bleeding episodes and by the rate of breakthrough bleeding during prophylaxis over ≥ 50 additional exposure days.
  Interventions: Biological: GreenGene™ F
- On-demand safety and efficacy substudy (Experimental): Hemostatic efficacy of GreenGene™ F will be assessed by its effectiveness in controlling spontaneous or traumatic bleeding episodes and by the rate of breakthrough bleeding in a minimum of 10 on demand treated subjects during additional 50 exposure days.
  Interventions: Biological: GreenGene™ F

INTERVENTIONS:
Biological: GreenGene™ F — Prophylaxis safety and efficacy substudy:
  intra venous infusion, 30 ± 10 IU/kg infusions 3 times per week with dose escalation to 45 ± 10 IU/kg if appropriate, for 50 exposure days
  Other Names: GreenGeneF; GreenGene F
  Arms: Prophylaxis safety and efficacy substudy
Biological: GreenGene™ F — On-demand safety and efficacy substudy:
  minor bleed = 20 ± 10 IU/kg moderate bleed = 30 ± 10 IU/kg major bleed = 30 - 50 IU/kg
  Other Names: GreenGeneF; GreenGene F
  Arms: On-demand safety and efficacy substudy

SUMMARY:
This study primarily will address the safety and secondarily will assess efficacy of GreenGene™ F in subjects with severe hemophilia A previously treated ≥50 exposure days with a GreenGene™ F, and without presence inhibitor to FVIII (Factor VIII).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have participated in the "GreenGene™ F_P3", (with Eudra CT number 2012-001445-40) or a pediatric study with GreenGene™ F
2. Have ≥50 previous exposure days to GreenGene™ F, as documented in the subject's medical records.
3. Negative assays for FVIII inhibitor at inclusion (<0.6BU Nijmegen assay), i.e. at the end of study "GreenGene™ F_P3" for patients entering into this extension study immediately after finishing the previous phase III study.
4. Normal liver and kidney function
5. Platelet count ≥ 100,000㎕
6. Normal prothrombin time or International Normalized Ratio (INR) < 1.5
7. Subjects receiving therapy for human immunodeficiency virus (HIV) or hepatitis must be on a stable treatment regimen
8. Subjects must be able to withhold FVIII infusions for approximately 72 h prior to each inhibitor assay
9. Absolute CD4 lymphocyte cell count ≥ 200㎕
10. Signed the written informed consent form or informed consent was obtained from the subject's legal guardian
11. Females must not be lactating or pregnant at screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [β-hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of β-hCG). A test was obtained more than 72 hours before the first dose of study drug
12. All females will be considered to be of childbearing potential unless they are appropriate age group and without other known or suspected cause) or have been sterilized surgically (i.e. bilateral tubal ligation, total hysterectomy or bilateral oophorectomy, all with surgery at least one month before dosing)
13. Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

1. Presence at Screening of FVIII inhibitor ≥ 0.6 BU as tested with the Nijmegen modification of the Bethesda assay.
2. Laboratory or clinical evidence of portal vein hypertension including, but not limited to, an INR > 1.4, the presence of splenomegaly and/or spider angiomata of physical examination and/or a history of esophageal hemorrhage or documented esophageal varices
3. Uncontrolled hypertension (diastolic blood pressure >100 mm Hg)
4. Hemoglobin < 10 g/dL
5. Severe renal dysfunction (creatinine > 2x upper limit of normal [ULN], total bilirubin > 2x the ULN)
6. Liver disease (alanine aminotransferase [ALT], aspartate aminotransferase [AST] > 3x the ULN)
7. History of diabetes or other metabolic disease
8. History of hypersensitivity or serious adverse reaction to recombinant or plasma-derived FVIII concentrates
9. History of pretreatment prior to the administration of FVIII products (e.g., antihistamines)
10. Regular use of antifibrinolytics or medications affecting platelet function
11. Hypersensitivity to hamster- or mouse derived proteins
12. Blood transfusions within 30 days of enrollment into the study
13. Current participation in another investigational drug or device study, or participated in a clinical study involving an investigational drug or device within 30 days of enrollment into the study
14. Unable or unwilling to cooperate with study procedures
15. Females who are pregnant (positive β-hCG test) or breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with development of inhibitors | every 3 months, up to 18 months
  Development of neutralizing antibodies (inhibitors) will be followed during the regular visits, average of 3 months.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Long Island Jewish Medical Center - Hemophilia Treatment Center, New Hyde Park, New York